CLINICAL TRIAL: NCT01378728
Title: Clinical Validation Study of a 'Hand-held' Point-of-Care Fluorescence Digital Imaging Device for Real-time Detection and Diagnosis of Wound Infections and Longitudinal Monitoring of Wound Healing Status
Brief Title: Clinical Validation of a 'Hand-held' Fluorescence Digital Imaging Device for Wound Care Applications
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: PRODIGI Wound Imaging Trial
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Wounds
Keywords: Optical imaging; Fluorescence imaging; Chronic and acute wounds; Wound bacteria; Bacterial biofilms; Pathogenic bacteria; Microorganisms; Wound infection; Wound healing; Treatment response assessment
MeSH Terms: conditions — Wounds and Injuries; Bronchiolitis Obliterans Syndrome; Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with chronic or acute wounds.: Patients with chronic or acute wounds.

SUMMARY:
The primary objective of this clinical study is to evaluate the use and effectiveness of our 'handheld' fluorescence digital imaging device platform for real-time non-invasive clinical monitoring of chronic wounds for healing and bacterial contamination/infectious status over time. This will enable us to determine if the device can detect and longitudinally track intrinsic changes that may occur during the wound healing process including, but not limited to, collagen re-modeling and bacterial infection of the wound site.

DETAILED DESCRIPTION:
Introduction and Rationale:

Wound care is a major clinical challenge and presents an enormous burden to health care worldwide. As wounds (chronic and acute) heal, a number of key biological changes occur at the wound site at the tissue and cellular level. Among these are inflammation, reformation of the epidermal barrier, and remodeling of the connective tissue in the dermis. However, a common major complication arising during the wound healing process, which can range from days to months, is bacterial infection. This can result in a serious impediment to the healing process and lead to significant complications, especially in chronic non-healing wounds. Currently, the standard wound care includes monitoring for possible infection by direct visual inspection under white light and by taking samples for analysis in the laboratory which takes approximately two days to provide a result. However, qualitative visual assessment only provides a gross view of the wound site (i.e., presence of purulent material and crusting) but does not provide the critically important information about underlying changes that are occurring at the tissue and cellular level (i.e., infection, matrix remodeling, inflammation, and necrosis).

All chronic wounds contain bacteria. But whether the wound is in bacterial balance (contamination with organisms on the surface or colonization with organisms in the tissue arranged in micro colonies without causing damage) or bacterial imbalance (critical colonization and infection) is of primary importance to healing. It is important to note that there is a continuum of bacterial presence pro¬gressing from bacterial balance to bacterial damage in a chronic wound. The diagnosis of infection is typically made clinically based on signs and symptoms in and around the local wound bed, the deeper structures, and the surrounding skin. The presence and severity of bacterial infection is typically diagnosed based on the clinical appearance of the wound under white light (i.e., pain, purulent exudate, crusting, swelling, erythema, heat). A major problem is that bacterial contamination within and around a wound cannot be determined directly by visualization of the bacteria themselves under white light, but is based on clinical signs and symptoms caused by bacterial contamination and/or infection within the wound (i.e., pain, purulent exudate, crusting, swelling, erythema, heat).

The remodeling and healing of connective tissues in wounds involves simultaneous synthesis and degradation of collagen fibrils. These bacteria include common species typically found at wound sites (i.e., Staphylococcus and Pseudomonas species). Bacterial swabs are collected at the time of wound examination and have the advantage of providing identification of specific bacterial/microbial species and quantification of bacterial burden. However, often, multiple swabs are collected randomly from the wound site and these are not targeted, and some swabbing techniques may spread the microorganisms around with the wound during the collection process, thus affecting patient healing time and morbidity. This may be a problem especially with large chronic (non-healing) wounds where the detection yield for bacterial presence is suboptimal, despite the collection of multiple swabs. Furthermore, bacteriological culture results often take about 2-4 days to come back from the laboratory, thus significantly delaying diagnosis and treatment. Thus, bacterial swabs do not provide real-time detection of infectious status of wounds. In addition, although wound swabbing appears to be straightforward, it can lead to inappropriate treatment, patient morbidity and increased hospital stays if not performed correctly. An image-based method that allows real-time monitoring of wound healing, particularly early dermal connective tissue remodeling, and the presence of bacterial contamination and/or infection over time could have a significant clinical impact.

Autofluorescence imaging has been used in gastroenterology to image both collagen and bacterial fluorescence in clinical studies. We wish to expand the use of tissue autofluorescence imaging technology to wound care and management in order to provide obtain biologically relevant information of the wound site at the tissue and biomolecular levels in real-time during the healing process. When used to assess wounds, tissue autofluorescence may aid in determining the degree of wound healing and the presence of bacterial infection. In preliminary preclinical testing, we have discovered that when wounds are illuminated a specific wavelength combination of excitation light, endogenous tissue components emit a characteristic fluorescent signal, while bacteria emit a unique fluorescence signal.

We have recently developed an innovative optical molecular imaging platform based on high-resolution fluorescence and white-light technologies in a hand-held, real-time, high-resolution, non-invasive (e.g. non-contact) format. This invention offers real-time detection of important biological and molecular information of a wound for the first time, and could have significant impact on improving conventional wound care and management. Based on extensive preclinical testing, the proposed technology has the capability of collecting autofluorescence images of wounds and detecting the presence and relative changes in connective tissue content and biodistribution involved in wound healing. It can also detect the earliest indication of bacterial/microorganism contamination within the wound (that are occult to standard white light visually-based assessment), thus providing a measure of infection status. This could significantly impact clinical wound care and management by i) reducing the complications associated with missed detection of bacteria infection, ii) facilitating image-guided swabbing/biopsy and iii) monitor wound healing over time. Furthermore, the compact and portable design of the imaging device platform makes it ideal for the clinical wound care environment as well as for point-of-care use for home-health care visits.

Study Objectives and Specific Aims

The primary objective of this clinical study is to evaluate the use and effectiveness of our 'handheld' fluorescence digital imaging device platform for real-time non-invasive clinical monitoring of chronic wounds for healing and bacterial contamination/infectious status over time. This will enable us to determine if the device can detect and longitudinally track intrinsic changes that may occur during the wound healing process including, but not limited to, collagen re-modeling and bacterial infection of the wound site.

As a secondary objective, we wish to obtain valuable end-user data on the clinical utility of the device within the wound clinic environment. This information will be used to optimize subsequent versions of the device during product development.

Most importantly, we hope to conclusively verify the added value that this imaging device brings to traditional wound care practice, and to what extent it will change the gold standard.

Specific Aims:

1. To determine if the fluorescence imaging device can detect changes in connective tissue over time that can be correlated with wound healing or re-modeling, compared with changes in wound size over time.
2. To determine the effectiveness of the fluorescence imaging device in detecting the presence (or contamination) of bacteria in and around a wound (including infection), compared with standard best practice methods (e.g. white light visualization and clinical signs and symptoms, with swabbing and bacteriology as the 'gold standard').
3. To identify the relationships between autofluorescence imaging of tissues and bacteria in wounds (including the wound margin) and the following: i) clinical signs of infection, ii) microbial load (i.e., number of organisms per gram of wound tissue), and iii) diversity of microbial species in the wound (i.e., number of different species isolated per wound), and Gram signing.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study according to the following criteria:

* > 18 years of age
* males and females
* presenting with chronic wounds (i.e., diabetic ulcers, etc.), with known or unknown infection status.

Exclusion Criteria:

Patients will be excluded in the study according to the following criteria:

* treatment with an investigational drug within 1 month before study enrolment
* any contra-indication to routine wound care and/or monitoring
* patients with pre-existing skin issues (e.g. melanomas, psoriasis) in areas close to wound(s) that will be studied
* inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients previously diagnosed with chronic and/or acute wounds will be considered for eligibility into this study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-02; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
wound size, bacterial load | 3 weeks after imaging with device

CONTACTS AND LOCATIONS:
Overall Officials: Ralph S DaCosta, PhD, Principal Investigator — Ontario Cancer Institute, University Health Network
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] DaCosta RS, Kulbatski I, Lindvere-Teene L, Starr D, Blackmore K, Silver JI, Opoku J, Wu YC, Medeiros PJ, Xu W, Xu L, Wilson BC, Rosen C, Linden R. Point-of-care autofluorescence imaging for real-time sampling and treatment guidance of bioburden in chronic wounds: first-in-human results. PLoS One. 2015 Mar 19;10(3):e0116623. doi: 10.1371/journal.pone.0116623. eCollection 2015. PMID 25790480